CLINICAL TRIAL: NCT03682393
Title: Does Post-operative Corticosteroid Treatment Prevent New-onset Atrial Fibrillation After Mitral Valve Surgery?
Brief Title: Post-operative Corticosteroid Treatment After Mitral Valve Surgery
Acronym: MitralPOCS
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: the study never started
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KUH5101126
Record Dates: First submitted 2018-09-18; First posted 2018-09-24 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Atrial Fibrillation
Keywords: postoperative; atrial fibrillation; post cardiac surgery; corticosteroid
MeSH Terms: conditions — Atrial Fibrillation | interventions — Hydrocortisone; Adrenal Cortex Hormones; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: half of the recruited patients will receive intravenous corticosteroid and the other half will receive intravenous isotonic saline as placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study is double blinded, neither the patients or investigators or nurses managing the drugs do not know whether the patient receives placebo (isotonic saline) or active drug (corticosteroid). In case of emergency the codes can be cracked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydrocortisone (Experimental): 100mg 1x3 hydrocortison intravenously for three days after mitral valve surgery or until atrial fibrillation onset
  Interventions: Drug: Hydrocortisone
- Placebos (Placebo Comparator): 100mg 1x3 intravenous fysiologic saline for three days after mitral valve surgery or until atrial fibrillation onset
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Hydrocortisone — 100mg 1x3 hydrocortison intravenously for three days after mitral valve surgery or until atrial fibrillation onset
  Other Names: corticosteroid
  Arms: Hydrocortisone
Drug: Placebos — 100mg 1x3 intravenous fysiologic saline for three days after mitral valve surgery or until atrial fibrillation onset
  Other Names: placebo, saline
  Arms: Placebos

SUMMARY:
The aim of the study is to intestigate whether three days intravenous corticosteroid management prevent atrial fibrillations in adults after mitral valve surgery. Prospective double-blinded randmized international multicenter study.

DETAILED DESCRIPTION:
Voluntary adult patients, who do not have persistent atrial fibrillation before mitral valve sugery will receive either intravenous corticosteroid or placebo on three postoperative days after mitral valve surgery. End points are atrial fibrillation onset or fullfilling the three days time limit. The study is double-blinded, randomized, prospective study and the aim is to recruite 240 patients. Patients are recruited from Oulu University Hospital, Finland, Kuopio University Hospital, Finland, Helsinki University Hospital, Finland, Turku University Hospital, Finland, Tampere Univerisity Hospital, Finland, Tartu University Hospital, Estonia, Tallinn Regionaalhaigla, Estonia and Liverpool Hospital, Sydney, Australia.

ELIGIBILITY:
Inclusion Criteria:

* open mitral valve surgery
* patients agrees to participate in the study
* adult (minimum 18 years of age)

Exclusion Criteria:

* atrial fibrillation onset before first postoperative morning
* prolonged intensive care unit stay (patient needs to stay in intensive care unit after first postoperative day)
* patient is underaged, does not want to participate or can not make the decision by himself or herself because of ie memory disability
* diabetes mellitus requiring insulin treatment and with recent hypo- or hyperglycemias which required hospital treatment
* systemic mucous infections
* known allergy or oversensitivity to hydrocortisone
* Cushing syndrome
* history of psychosis
* history of ulcus or active ulcus
* chronic atrial fibrillation or atrial flutter
* corticosteroid or immunosuppressive treatment in use for any reason
* active tuberculosis infection
* severe renal impairment (serum creatinine 200 umol/l or over)
* history of deep or superficial venous trombosis
* Herpes simplex -ceratitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
atrial fibrillation | three days after mitral valve surgery
  Atrial fibrillation onset in the timeframe of three postoperative days after mitral valve surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jari Halonen, MD, PhD, Principal Investigator — general surgery attending, clinical teacher
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No
IPD are not to be shared with other researchers.